CLINICAL TRIAL: NCT00385281
Title: Proteomic Profiling for Influenza Vaccination, 2nd Study: FluMist
Brief Title: Proteomic Profiling for Influenza Vaccination - FluMist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06-0041
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-03

CONDITIONS: Influenza
Keywords: proteomic profiling, influenza, vaccine, FluMist
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

INTERVENTIONS:
Biological: FluMist

SUMMARY:
The purpose of this study is to look at changes that occur in blood and nasal swab samples after a person's immune system responds to receiving a flu vaccine. The investigators will look at the immune response in 50 healthy volunteers, between 21 and 49 years of age, after they have been vaccinated with 1 dose of a flu vaccine sprayed into the nose. A blood sample and nasal swab of each nostril will be collected from volunteers before they receive the flu vaccination. After receiving the flu vaccine, volunteers will record health changes and daily temperatures on diary cards at home for 21 days. Blood will be drawn and nasal swabs will be collected from each volunteer at each of the 6 study visits. Volunteers will participate in the study for approximately 1 month. This study is being conducted at the Glennan Center for Geriatrics and Gerontology at Eastern Virginia Medical School.

DETAILED DESCRIPTION:
This is a nonrandomized, non-comparative study conducted in 50 healthy subjects, between 21 and 49 years of age, who have been vaccinated with 1 dose (0.5 mL) of Influenza Virus Vaccine Live, Intranasal FluMistTM, a live trivalent nasally administered vaccine. The central hypothesis is that immune responses to vaccination can be quantified by proteomic profiling of serum and nasal proteins, and that host responses to different infectious agents are unique and can be "fingerprinted" by proteomics. Using influenza virus vaccination, this study proposes to use mass spectrometry platforms to profile and characterize proteins from serum samples obtained from recipients. These samples will be used to develop a proteomic profiling system for monitoring vaccine response, and will eventually allow earlier detection/diagnosis of infection. Annually, natural influenza infections cause serious international public health problems that are particularly severe in elderly people, who account for more than 90% of influenza mortality. The current trivalent split virus influenza vaccine is cost-effective, but its efficacy is greatly reduced in the elderly population. The long-term goal of the investigators' approach is to develop tools useful for reducing the morbidity and mortality of influenza from natural and potential bioterrorism-related infections by improving measures of vaccine efficacy and early diagnosis. This study is being conducted at the Glennan Center for Geriatrics and Gerontology at Eastern Virginia Medical School. Solicited adverse events (AEs) and daily temperatures will be collected on diary cards for 21 days. Unsolicited AEs will also be collected throughout the duration of the study. Blood will be drawn and nasal swabs will be collected from each subject at each of the 6 study visits. Subjects will participate in the study for approximately 1 month. The primary objective of this study is to analyze serum samples before and after FluMist intranasal attenuated live-virus influenza vaccination to identify surrogate markers reflective of the immune response by using surface-enhanced laser desorption/ionization-time of flight (SELDI-TOF) and matrix-assisted laser desorption/ionization-time of flight (MALDI-TOF) mass spectrometry proteomic profiling tools reflective of the immune response. Concurrent T-cell activation, cytokine assays, and hemagglutination inhibition (HI) serologic assays will correlate cellular and humoral responses to influenza vaccination with protein profiling changes. Proteins obtained from intranasal swabs pre and post vaccination will be analyzed. The investigators anticipate identifying multiple host response proteins from this analysis using combinations of gel electrophoresis, MALDI-TOF and tandem MS/MS approaches. The secondary objective is safety. Data on solicited reactions will be collected from Day 0 to Day 14. The time of occurrence of AEs will be used to determine if there is a correlation with the time of increase in certain protein biomarkers. The primary endpoint is to identify surrogate markers reflective of the immune response in serum and/or nasal proteins and to correlate these markers to cellular and humoral responses (demonstrated with T-cell activation, cytokine assays, and the hemagglutination inhibition [HI] serologic assays) to influenza vaccination. The secondary endpoint is safety. Data on local reactions and solicited systemic reactions will be collected from Day 0 to Day 14 and categorized according to severity. Unsolicited AEs will be collected and categorized throughout the study by severity, duration, and relatedness to vaccine. The time of occurrence of AEs will be used to determine if there is a correlation with the time of increase in certain protein biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages of 21 to 49 years of age on day of enrollment, visit 1(day 0).
2. Provides written informed consent.
3. Subject is judged to be healthy on the basis of verbal medical and concomitant medications history and has been medically stable prior to screening
4. Subject is able to attend scheduled visits and to comply with the study procedures during the entire duration of the study and will be available for 1 month after enrollment.
5. Female is not at risk of pregnancy, based on the following:

   1. Utilizing adequate method of birth control and agree to continue using this method for at least 1 month after enrollment. Adequate methods of birth control may include hormonal (oral, transdermal, or injectable) or double barrier methods (eg condom with spermicide, vaginal combined ring) or intra-uterine device. If using hormonal method or intra-uterine device, usage should be stable for 1 month prior to vaccination and should continue for 1 month post vaccination.
   2. Negative urine pregnancy test is required for all females at study entry. Females surgically sterilized (history of tubal ligation or total or subtotal hysterectomy) or post-menopausal for 2 years must still have a negative pregnancy test at time of enrollment.
6. Subject should be available through telephone contact and agree to participate in all scheduled visits.

Exclusion Criteria:

1. Adults younger than 21 years of age or 50 years and older
2. Subject had physician-diagnosed (preferably by culture) influenza at any time during the past 2 years.
3. Subject received an influenza vaccine in the 6 months preceding enrollment in the study
4. Subjects who receive any live virus vaccine within one month of enrollment and any inactivated or subunit vaccine within 2 weeks of enrollment or with plans to receive any vaccine during this study will be excluded from the study, eg, pneumococcal vaccine.
5. Subject received blood or blood products in the last 3 months.
6. Subject has asthma or reactive airway disease.
7. Subject has a history of any serious vaccine reactions or anaphylaxis or reactions likely to be exacerbated by any component of the study vaccine,
8. Subject is allergic to eggs, egg products or gentamycin.
9. Subject has known or suspected disease(s) of the immune system with immunosuppression, eg, rheumatoid arthritis, systemic lupus erythematosus (SLE), lymphoma, human immunodeficiency virus (HIV), cancer diagnoses or treatment within the last 5 years (except skin cancer), etc.
10. Subject is currently being treated with an immunosuppressive medications (ie, cancer therapeutic agents such as tamoxifen, systemic corticosteroids such as prednisone, and arthritis medications such as methotrexate). Please note that inhaled or topical corticosteriods are acceptable.
11. FluMist recipients in close contact (eg, within the same household) with immunocompromised individuals during periods in which the immunosuppressed person requires care in a protective environment. (contact should be avoided for at least 21 days). Contact with small children is not an exclusion. Females who breastfeed are excluded.
12. Drug interactions: On antiviral therapy in 48 hours preceding scheduled vaccination
13. Antiviral agents administered until 3 weeks after FluMist vaccination.
14. Participation in any other interventional drug or vaccine trial within 30 days prior to enrollment. Therefore subject is not to receive other investigational products (drug or vaccine) during the length of their participation in the trial.
15. Subject has acute respiratory illness. Administration of FluMist should be postponed until after the acute phase (at least 72 hours) of respiratory illnesses.
16. Subject has active infections or illnesses.
17. Subject had an acute illness with or without fever (temperature >/= 99.5 F [oral]) in the 72 hours preceding vaccination. Administration of FluMist should be postponed until after the acute phase (at least 72 hours) of febrile and/or acute illnesses.
18. Subject has acute or chronic medical health condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include, but are not limited to health problems associated with

    1. heart disease, (if heart failure is present, New York Heart Association Functional Class III or IV),
    2. kidney disease, (history of significant renal impairment e.g., dialysis and treatment for kidney disease, including diabetic and hypertensive kidney disease),
    3. chronic liver disorders (e.g. hepatitis B or C),
    4. diabetes mellitus (excluding diet-controlled diabetes),
    5. arteriosclerotic event during the 6 months prior to enrollment (eg, history of myocardial infarction, stroke, recanalization of femoral arteries, or transient ischemic attack),
    6. functional or anatomic asplenia,
    7. cancer diagnosed and treated within the past 5 years with chemotherapy, radiation therapy and/or surgery
    8. significant anemia or other blood disorders.
    9. Underlying unstable chronic disease e.g.uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg at Visit 1), etc.
19. Subject has any active neurologic disorders (ie, encephalopathy, optic neuritis/neuropathy, partial facial paralysis, and brachial plexus neuropathy).
20. Subject is pregnant or planning to become pregnant within the next 2 months.
21. Subject is breastfeeding.
22. Subject has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
23. Subject has a prior history of Guillain-Barré syndrome.
24. Subject has a history of drug or alcohol abuse.

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States